CLINICAL TRIAL: NCT03449030
Title: An Open-Label, Dose Escalation, Phase 1, First-in-Human Study of TAK-164, an Antibody-Drug Conjugate, in Patients With Advanced Gastrointestinal Cancers Expressing Guanylyl Cyclase C
Brief Title: A Study of TAK-164 in Participants With Advanced Gastrointestinal (GI) Cancer Expressing Guanylyl Cyclase C (GCC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient clinical benefit to participants at the selected recommended phase 2 (RP2D) dose in Part A.
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: TAK-164-1001; U1111-1207-9923 (Other: WHO); 2018-002214-12 (Registry Identifier: EudraCT)
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Results first posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-02

CONDITIONS: Gastrointestinal Neoplasms; Esophageal, Stomach, Pancreas, Colon Neoplasms; Malignant Tumors of Digestive Organ; Advanced Gastrointestinal Malignancies
Keywords: Drug Therapy
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A Escalation Stage: TAK-164 Q3W (Experimental): TAK-164 0.004 milligram per kilogram (mg/kg) starting dose, intravenous infusion, until PD, unacceptable toxicity or discontinuation by participant. Dose escalation will be performed to determine the MTD and/or RP2D.
  Interventions: Drug: TAK-164
- Part B Expansion Stage: TAK-164 Q3W (Experimental): TAK-164, intravenous infusion, until PD, unacceptable toxicity or discontinuation by participant. TAK-164 RP2D dose to be decided based on safety, PK, pharmacodynamics and antitumor response data observed in Part A escalation stage.
  Interventions: Drug: TAK-164
- Part C Imaging Substudy: 89Zr-TAK-164 and TAK-164 (Experimental): 89Zr-TAK-164, intravenous infusion, followed by unlabeled TAK-164, intravenous infusion in combination with 89Zr-TAK-164, intravenous infusion, and further followed by unlabeled TAK-164, intravenous infusion, until PD, unacceptable toxicity or discontinuation by participant. TAK-164 recommended imaging dose (RID) or RP2D dose to be decided based on safety, PK, PD and antitumor response data observed in Part A escalation stage.
  Interventions: Drug: TAK-164; Drug: 89Zr-TAK-164

INTERVENTIONS:
Drug: TAK-164 — TAK-164 intravenous infusion.
Drug: 89Zr-TAK-164 — 89Zr-TAK-164 intravenous infusion
  Arms: Part C Imaging Substudy: 89Zr-TAK-164 and TAK-164

SUMMARY:
The purpose of this study is to evaluate the safety of TAK-164 and to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) and schedule.

DETAILED DESCRIPTION:
The drug being tested in this study is a novel antibody-drug conjugate (ADC) called TAK-164. TAK-164 is being evaluated in participants with advanced GCC-positive GI cancer (Part A) or colorectal carcinoma (CRC) and gastric carcinoma (Part B and Part C) to determine safety, tolerability, and pharmacokinetics (PK) and MTD/RP2D of TAK-164, as well as the preliminary efficacy. The study will include approximately 100 evaluable participants.

In Part A (Escalation), approximately 25 participants with GI carcinoma will be enrolled. Those include participants with various GI malignancies such as carcinomas of esophagus, stomach, colon, and pancreas. The starting dose for Arm 1 will be 0.004 mg/kg of TAK-164 administered intravenously on Day 1 Q3W and the maximal dose will not exceed 0.19 mg/kg Q3W.

In Part B (Expansion), approximately 50 participants will be enrolled to receive TAK-164 infusion at determined RP2D in Part A. Participants will follow the Q3W schedule and will be followed until PD, unacceptable toxicity, or until they choose to withdraw consent.

In Part C (Imaging substudy to be conducted in the Netherlands only), approximately 25 participants with GCC-expressing metastatic colorectal carcinoma (mCRC) will be enrolled to receive 89Zr-TAK-164 and unlabeled TAK-164 at determined RP2D in Part A.

This multi-center trial will be conducted in the United States and the Netherlands. The overall time to participate in this study is up to 55 months. Participants will attend an end of study (EOS) visit 30 days after the last dose of TAK-164 or just prior to the start of subsequent antineoplastic therapy, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed measurable advanced and/or metastatic solid GI tumor that expresses GCC protein (H-score greater than or equal to [>=] 10), for which standard treatment is no longer effective or does not offer curative or life-prolonging benefit. For the escalation part of the study (Part A), GI malignancies include, but are not limited to, metastatic colorectal carcinoma (mCRC), gastric carcinoma, esophageal carcinoma, small intestine cancer, and pancreatic cancer. The expansion part of the study (Part B) is limited to participants with CRC expressing a high-level of GCC (H-Score >=150) and gastric carcinoma (H-Score >=10). Part C includes participants with CRC and gastric carcinoma (H-score >=10 for both indications).

   o Part B of the study will be limited to participants with 2 or 3 prior lines of systemic standard of care therapy.
2. Male or female participants 18 years or older.
3. Adequate bone marrow function, defined as an absolute neutrophil count (ANC) of >=1.5*10^9 per liter (/L), platelet count >=100*10^9/L, and hemoglobin >=9 gram per deciliter (g/dL). Receiving transfusions or hematopoietic growth factors to meet enrollment criteria is not allowed within 14 days preceding the first dose of study drug.
4. Adequate hepatic function with total bilirubin less than or equal to (<=) 1.5* upper limit of normal (ULN), serum ALT and AST must be less than (<) 2.5*ULN (AST and ALT may be elevated up to 3*ULN if the elevation can be reasonably ascribed to the presence of metastatic disease in liver), serum albumin > 3.0 g/dL.
5. Adequate renal function as defined by creatinine CL >= 60 milliliter per minute (mL/min).
6. Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1.
7. Life expectancy of at least 12 weeks.
8. Completion of prior chemotherapy, biologic therapy, immunotherapy, or radiation therapy at least 4 weeks prior to enrollment.
9. Resolution of all toxic effects of prior treatments (except alopecia) to Grade <=1 NCI CTCAE, version 5.
10. A portion of participants should have tumors amenable for serial biopsy and a willingness to provide consent for pharmacodynamic assessment.

    Additionally for Part C (imaging sub study), participant must fulfill the following criteria:
11. At least 1 extrahepatic metastatic lesion >=2 centimeter (cm) in the longest diameter.

Exclusion Criteria:

1. Treatment with anticancer chemotherapy or biologic therapy or with an experimental anticancer agent within 28 days of the initial dose of study drug.
2. Diagnosed or treated for another malignancy within 2 years before administration of the first dose of study drug, or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
3. Participant has a history of severe allergic or anaphylactic reactions to recombinant proteins or excipients used in TAK-164 formulation or 89Zr-TAK-164 formulation.
4. Use of strong cytochrome P3A (CYP3A) inhibitors and CYP3A inducers or inhibitors or modulators of P-glycoprotein (P-gp) or breast cancer resistance protein (BCRP) within 1 week before the first dose of study drug.
5. For participants enrolled in studies in which tumor biopsies are obtained:

   * Known bleeding diathesis or history of abnormal bleeding, or any other known coagulation abnormalities that would contraindicate the tumor biopsy procedure.
   * Ongoing therapy with any anticoagulant or antiplatelet agents (example, aspirin, clopidogrel, heparin, or warfarin).
6. Participant has concurrent alcohol abuse or a history of drug-induced liver injury (DILI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - SCRI - Tennessee Oncology Nashville - Southern Hills Clinic, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Kim R, Leal AD, Parikh A, Ryan DP, Wang S, Bahamon B, Gupta N, Moss A, Pye J, Miao H, Inguilizian H, Cleary JM. A phase I, first-in-human study of TAK-164, an antibody-drug conjugate, in patients with advanced gastrointestinal cancers expressing guanylyl cyclase C. Cancer Chemother Pharmacol. 2023 Apr;91(4):291-300. doi: 10.1007/s00280-023-04507-w. Epub 2023 Feb 4. PMID 36738333
- [Derived] Abu-Yousif AO, Cvet D, Gallery M, Bannerman BM, Ganno ML, Smith MD, Lai KC, Keating TA, Stringer B, Kamali A, Eng K, Koseoglu S, Zhu A, Xia CQ, Landen MS, Borland M, Robertson R, Bolleddula J, Qian MG, Fretland J, Veiby OP. Preclinical Antitumor Activity and Biodistribution of a Novel Anti-GCC Antibody-Drug Conjugate in Patient-derived Xenografts. Mol Cancer Ther. 2020 Oct;19(10):2079-2088. doi: 10.1158/1535-7163.MCT-19-1102. Epub 2020 Aug 11. PMID 32788205

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in the United States from 23 April 2018 to 27 February 2020.
Pre-assignment Details: Participants with advanced gastrointestinal (GI) cancers expressing guanylyl cyclase C (GCC) were enrolled in this study to receive TAK-164, every 3 weeks in Part A (Dose Escalation) of the study. Study was terminated after completion of Part A and prior to start of Parts B (Expansion Cohort) and C (Imaging Substudy) because there was insufficient clinical benefit to participants at the selected recommended phase 2 (RP2D) dose in Part A.
Groups:
- Part A: TAK-164 0.004 mg/kg: TAK-164 0.004 milligram per kilogram (mg/kg), intravenous infusion, on Day 1 of each 21-day treatment cycle until progressive disease (PD), unacceptable toxicity or discontinuation by participant.
- Part A: TAK-164 0.008 mg/kg: TAK-164 0.008 mg/kg, intravenous infusion, on Day 1 of each 21-day treatment cycle until PD, unacceptable toxicity or discontinuation by participant.
- Part A: TAK-164 0.016 mg/kg: TAK-164 0.016 mg/kg, intravenous infusion, on Day 1 of each 21-day treatment cycle until PD, unacceptable toxicity or discontinuation by participant.
- Part A: TAK-164 0.032 mg/kg: TAK-164 0.032 mg/kg, intravenous infusion, on Day 1 of each 21-day treatment cycle until PD, unacceptable toxicity or discontinuation by participant.
- Part A: TAK-164 0.064 mg/kg: TAK-164 0.064 mg/kg, intravenous infusion, on Day 1 of each 21-day treatment cycle until PD, unacceptable toxicity or discontinuation by participant.
- Part A: TAK-164 0.12 mg/kg: TAK-164 0.12 mg/kg, intravenous infusion, on Day 1 of each 21-day treatment cycle until PD, unacceptable toxicity or discontinuation by participant.
- Part A: TAK-164 0.16 mg/kg: TAK-164 0.16 mg/kg, intravenous infusion, on Day 1 of each 21-day treatment cycle until PD, unacceptable toxicity or discontinuation by participant.
- Part A: TAK-164 0.19 mg/kg: TAK-164 0.19 mg/kg, intravenous infusion, on Day 1 of each 21-day treatment cycle until PD, unacceptable toxicity or discontinuation by participant.
- Part A: TAK-164 0.25 mg/kg: TAK-164 0.25 mg/kg, intravenous infusion, on Day 1 of each 21-day treatment cycle until PD, unacceptable toxicity or discontinuation by participant.
- Part A: TAK-164 0.32 mg/kg: TAK-164 0.32 mg/kg, intravenous infusion, on Day 1 of each 21-day treatment cycle until PD, unacceptable toxicity or discontinuation by participant.
Period: Overall Study
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Started | 1 | 1 | 1 | 5 | 7 | 7 | 2 | 3 | 3 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 5 | 7 | 7 | 2 | 3 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 0
Not completed — Symptomatic Deterioration | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Not completed — Progressive Disease | 1 | 0 | 1 | 4 | 5 | 3 | 0 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population was defined as all participants who received at least 1 dose of study drug.
Groups:
- Part A: TAK-164 0.004 mg/kg: TAK-164 0.004 mg/kg, intravenous infusion, on Day 1 of each 21-day treatment cycle until PD, unacceptable toxicity or discontinuation by participant.
- Total: Total of all reporting groups
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg | Total
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 7 | 7 | 2 | 3 | 3 | 1 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (NA) — Standard deviation could not be calculated because only one participant was evaluable. | 52.0 (NA) — Standard deviation could not be calculated because only one participant was evaluable. | 59.0 (NA) — Standard deviation could not be calculated because only one participant was evaluable. | 55.2 (8.14) | 57.1 (8.36) | 48.0 (13.11) | 53.0 (14.14) | 65.3 (3.21) | 48.0 (3.61) | 39.0 (NA) — Standard deviation could not be calculated because only one participant was evaluable. | 54.2 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 4 | 4 | 4 | 1 | 1 | 0 | 1 | 18
  Male | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 2 | 3 | 0 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 1 | 4 | 6 | 7 | 2 | 3 | 3 | 1 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  White | 1 | 1 | 1 | 4 | 6 | 5 | 2 | 2 | 3 | 0 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 1 | 5 | 7 | 7 | 2 | 3 | 3 | 1 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLTs were evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5. DLT was defined as any of the following adverse events (AEs) that occurred and were considered by the investigator to be related to therapy with study drug: hematologic toxicities were, Grade 4 neutropenia (absolute neutrophil count [ANC] less than (<) 500 cells/cubic millimeter [mm^3]), thrombocytopenia (platelets <25,000/mm^3), febrile neutropenia (ANC <1000/mm^3) with fever (greater than [>] 38.3 degree Celsius or sustained temperature of greater than or equal to (>=) 38 degree Celsius, Grade 3 or greater thrombocytopenia with clinically meaningful bleeding at any time, Grade 3 or greater nausea and/or emesis that occurs despite the use of optimal anti-emetic prophylaxis and Grade 3 or greater diarrhea that occurs despite optimal supportive care measures and any other Grade 3 or greater nonhematologic toxicity except brief (<1 week) Grade 3 fatigue.
Time Frame: Baseline up to Month 22
Population: The safety population was defined as all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 7 | 7 | 2 | 3 | 3 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0

2. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: From first dose of study drug up to 30 days following the last dose of study drug (up to 22 months)
Population: The safety population was defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 7 | 7 | 2 | 3 | 3 | 1
percentage of participants | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100

3. Primary Outcome: Percentage of Participants With Grade 3 or Above AEs
Description: AE Grades were evaluated as per NCI CTCAE, version 5. Graded from Grade 1: Mild asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated, Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL), Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL, Grade 4: Life-threatening consequences; urgent intervention indicated, Grade 5: Death related AE. Higher grade indicates more severe condition.
Time Frame: From first dose of study drug up to 30 days following the last dose of study drug (up to 22 months)
Population: The safety population was defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 7 | 7 | 2 | 3 | 3 | 1
percentage of participants | 0 | 100 | 100 | 60 | 14.3 | 71.4 | 50.0 | 100 | 100 | 0

4. Primary Outcome: Percentage of Participants With Drug-related AEs
Time Frame: From first dose of study drug up to 30 days following the last dose of study drug (up to 22 months)
Population: The safety population was defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 7 | 7 | 2 | 3 | 3 | 1
percentage of participants | 100 | 0 | 100 | 100 | 85.7 | 71.4 | 50.0 | 66.7 | 66.7 | 100

5. Primary Outcome: Percentage of Participants With Drug-related Grade 3 or Above AEs
Description: AE Grades were evaluated as per NCI CTCAE, version 5. Graded from Grade 1: mild asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated, Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL, Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL, Grade 4: Life-threatening consequences; urgent intervention indicated, Grade 5: death related AE. Higher grade indicates more severe condition.
Time Frame: From first dose of study drug up to 30 days following the last dose of study drug (up to 22 months)
Population: The safety population was defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 7 | 7 | 2 | 3 | 3 | 1
percentage of participants | 0 | 0 | 100 | 20.0 | 14.3 | 42.9 | 50.0 | 33.3 | 66.7 | 0

6. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Time Frame: From first dose of study drug up to 30 days following the last dose of study drug (up to 22 months)
Population: The safety population was defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 7 | 7 | 2 | 3 | 3 | 1
percentage of participants | 0 | 100 | 0 | 60 | 0 | 42.9 | 50.0 | 66.7 | 66.7 | 0

7. Primary Outcome: Percentage of Participants With AEs Leading to Discontinuation
Time Frame: From first dose of study drug up to 30 days following the last dose of study drug (up to 22 months)
Population: The safety population was defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 7 | 7 | 2 | 3 | 3 | 1
percentage of participants | 0 | 0 | 0 | 0 | 0 | 28.6 | 0 | 0 | 33.3 | 0

8. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-164
Time Frame: Cycles 1 and 2 Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose (Cycle length = 21 days)
Population: Pharmacokinetic (PK) analysis was not conducted due to premature discontinuation of the study after completion of Part A and prior to start of Parts B (Expansion Cohort) and C (Imaging Substudy) because there was insufficient clinical benefit to participants at the selected RP2D dose in Part A.
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Tmax: Time to Reach the Maximum Observed Plasma Concentration (Cmax) for TAK-164
Time Frame: Cycles 1 and 2 Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose (Cycle length = 21 days)
Population: PK analysis was not conducted due to premature discontinuation of the study after completion of Part A and prior to start of Parts B (Expansion Cohort) and C (Imaging Substudy) because there was insufficient clinical benefit to participants at the selected RP2D dose in Part A.
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to Time of Last Quantifiable Concentration for TAK-164
Time Frame: Cycles 1 and 2 Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose (Cycle length = 21 days)
Population: as for outcome 9
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Ctrough: Observed Concentration Measured at the End of a Dosing Interval for TAK-164
Time Frame: Cycles 1 and 2 Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose (Cycle length = 21 days)
Population: as for outcome 9
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was assessed by the investigator based on modified Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. ORR was defined as the percentage of participants who had complete response (CR) or partial response (PR). CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to <10 millimeters (mm). PR was defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum longest diameter.
Time Frame: From start of study treatment until the start of subsequent anti cancer therapy ( up to Month 22)
Population: The response-evaluable population was defined as participants who received at least 1 dose of study drug, had measurable disease at baseline, and had at least 1 post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 6 | 5 | 2 | 2 | 1 | 1
percentage of participants | 0 [0.0 to 97.5] | 100 [2.5 to 100.0] | 0 [0.0 to 97.5] | 0 [0.0 to 52.2] | 0 [0.0 to 45.9] | 0 [0.0 to 52.2] | 0 [0.0 to 84.2] | 0 [0.0 to 84.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]

13. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with CR, PR or stable disease (SD). DCR was assessed based on modified RECIST version 1.1 criteria. CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since the treatment started.
Time Frame: Baseline up to Month 22
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 6 | 5 | 2 | 2 | 1 | 1
percentage of participants | 100 [2.5 to 100.0] | 100 [2.5 to 100.0] | 100 [2.5 to 100.0] | 40.0 [5.3 to 85.3] | 50.0 [11.8 to 88.2] | 40.0 [5.3 to 85.3] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]

14. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first documentation of a response (CR or PR) to the date of first documented PD or death due to any cause, whichever occurred first based on modified RECIST version 1.1 criteria. CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum longest diameters. PD was >=20% increase in sum of diameters of target lesions, reference-smallest sum recorded in study (sum at baseline if that was smallest). Sum of diameters must have absolute increase of >=5 mm. Appearance of >=1 new lesions also considered PD.
Time Frame: From the date of first documentation of a response (CR or PR) to the date of first documented PD or death due to any cause, whichever occurred first (up to 22 months)
Population: The response-evaluable population was defined as participants who received at least 1 dose of study drug, had measurable disease at baseline, and had at least 1 post-baseline disease assessment. Here 'N' (Overall number of participants analyzed) signifies participants with events CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
months |  | NA [NA to NA] — Median, lower and upper limit of 95% CI could not be calculated because none of the participant had an event (PD or death) |  |  |  |  |  |  |  |

15. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from date of first study drug administration to the day of first documented PD or death due to any cause, whichever occurred first according to modified RECIST version 1.1 criteria. PD was >= 20% increase in sum of diameters of target lesions, reference-smallest sum recorded in study (sum at baseline if that was smallest). Sum of diameters must have absolute increase of >=5 mm. Appearance of >=1 new lesions also considered PD. PFS was censored at the last response assessment that is stable disease or better, prior to receipt of subsequent anticancer therapy, if applicable. Participants with no post-baseline assessments was censored at Day 1.
Time Frame: From date of first study drug administration to the day of first documented PD or death due to any cause, whichever occurred first (up to 22 months)
Population: The response-evaluable population was defined as participants who received at least 1 dose of study drug, had measurable disease at baseline, and had at least 1 post-baseline disease assessment. Here 'N' (Overall number of participants analyzed) signifies participants with events (PD or/and death).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Number analyzed (Participants) | 1 | 0 | 1 | 4 | 6 | 3 | 1 | 2 | 1 | 1
months | 2.79 [NA to NA] — Lower and upper limit of 95% CI could not be calculated because only one participant had an event. |  | 6.24 [NA to NA] — Lower and upper limit of 95% CI could not be calculated because only one participant had an event. | 1.35 [0.59 to NA] — Upper limit of 95% CI could not be calculated because insufficient number of participants had an event. | 1.91 [1.22 to 3.48] | 1.58 [1.08 to 1.58] | 1.41 [NA to NA] — Lower and upper limit of 95% CI could not be calculated because only one participant had an event. | 1.81 [1.25 to 2.37] | 1.05 [NA to NA] — Lower and upper limit of 95% CI could not be calculated because only one participant had an event. | 1.18 [NA to NA] — Lower and upper limit of 95% CI could not be calculated because only one participant had an event.

16. Secondary Outcome: Number of Participants With Positive Antidrug Antibody (ADA) Levels in Serum
Time Frame: Baseline up to Month 22
Population: The immunogenicity evaluable population was defined as all participants with a baseline immunogenicity assessment and at least 1 postbaseline immunogenicity assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 7 | 6 | 2 | 1 | 3 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

17. Primary Outcome: Recommended Phase 2 Dose (RP2D) of TAK-164
Description: RP2D was the highest safe dose that could be applied to the expansion phase.
Time Frame: Baseline up to Month 22
Population: The safety population was defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: mg/kg
Groups:
- Part A: TAK-164: TAK-164 0.004, 0.008, 0.016, 0.032, 0.064, 0.12, 0.16, 0.19, 0.25 or 0.32 mg/kg, intravenous infusion, on Day 1 of each 21-day treatment cycle until PD, unacceptable toxicity or discontinuation by participant.
Arm/Group | Part A: TAK-164
Number analyzed (Participants) | 31
mg/kg | 0.064

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug up to 30 days following the last dose of study drug (up to 22 months)
Description: At each visit the investigator had to assess any occurrence of adverse events. Participants may report adverse events occurring at any other time during the study. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety data for markedly abnormal values for laboratory tests and vital sign are embedded in this AE section.
Arm/Group | Part A: TAK-164 0.004 mg/kg | Part A: TAK-164 0.008 mg/kg | Part A: TAK-164 0.016 mg/kg | Part A: TAK-164 0.032 mg/kg | Part A: TAK-164 0.064 mg/kg | Part A: TAK-164 0.12 mg/kg | Part A: TAK-164 0.16 mg/kg | Part A: TAK-164 0.19 mg/kg | Part A: TAK-164 0.25 mg/kg | Part A: TAK-164 0.32 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/5 | 1/7 | 0/7 | 0/2 | 1/3 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 0/1 | 3/5 | 0/7 | 3/7 | 1/2 | 2/3 | 2/3 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 5/5 | 7/7 | 6/7 | 2/2 | 3/3 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: TAK-164 0.004 mg/kg (N=1) | Part A: TAK-164 0.008 mg/kg (N=1) | Part A: TAK-164 0.016 mg/kg (N=1) | Part A: TAK-164 0.032 mg/kg (N=5) | Part A: TAK-164 0.064 mg/kg (N=7) | Part A: TAK-164 0.12 mg/kg (N=7) | Part A: TAK-164 0.16 mg/kg (N=2) | Part A: TAK-164 0.19 mg/kg (N=3) | Part A: TAK-164 0.25 mg/kg (N=3) | Part A: TAK-164 0.32 mg/kg (N=1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: TAK-164 0.004 mg/kg (N=1) | Part A: TAK-164 0.008 mg/kg (N=1) | Part A: TAK-164 0.016 mg/kg (N=1) | Part A: TAK-164 0.032 mg/kg (N=5) | Part A: TAK-164 0.064 mg/kg (N=7) | Part A: TAK-164 0.12 mg/kg (N=7) | Part A: TAK-164 0.16 mg/kg (N=2) | Part A: TAK-164 0.19 mg/kg (N=3) | Part A: TAK-164 0.25 mg/kg (N=3) | Part A: TAK-164 0.32 mg/kg (N=1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 3 (4) | 1 (1) | 1 (2) | 0 (0) | 2 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 4 (5) | 3 (5) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (4) | 5 (6) | 3 (3) | 5 (11) | 1 (1) | 1 (3) | 3 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 4 (6) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 3 (5) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 3 (3) | 1 (2) | 1 (1) | 2 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder discomfort (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0)
Skin swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT03449030/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT03449030/SAP_001.pdf